CLINICAL TRIAL: NCT04743089
Title: Cost-Effectiveness of Spyglass Direct Visualization System Facilitated Management for the Patients With Intrahepatic Bile Duct Stone and/or Large Extrahepatic Bile Duct Stone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2018-0031
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Patients With Large or Impacted Intra- or Extra-hepatic Bile Duct Stone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spyglass arm (Experimental): Patients who underwent IHD/EHD stone removal by ERCP with SpyGlass™ DS Direct Visualization System.
  Interventions: Device: ERCP using SpyGlass™ DS Direct Visualization System
- PTCS arm (historical cohort) (Other): Patients who underwent IHD/EHD stone removal by PTCS
  Interventions: Other: PTCS

INTERVENTIONS:
Device: ERCP using SpyGlass™ DS Direct Visualization System — Lithotripsy and stone removal will be performed using ERCP and Spyglass system to patients with IHD/EHD stone, which is difficult to remove through conventional ERCP. The SpyGlass™ DS Direct Visualization System will be applied directly into the bile duct via the working channel of the duodenoscope. Under the high-resolution digital imaging, lithotripsy such as EHL could be done.
  Arms: Spyglass arm
Other: PTCS — A historical cohort of patients who underwent PTCS to remove bile duct stones which is difficult to treat by ERCP.
  Arms: PTCS arm (historical cohort)

SUMMARY:
Endoscopic retrograde cholangio-pancreatectomy (ERCP) is the most commonly used endoscopic method for the treatment of biliary diseases including choledocholithiasis. When the ERCP cannot be performed under fluoroscopy due to various reasons such as the location of disease (i.e. intrahepatic bile duct lesion) and characteristics of the bile duct (i.e. altered anatomy, stenosis etc.), percutaneous transhepatic cholangiography (PTCS) is performed as an another treatment option. However, treatment of biliary lesions via PTCS requires at least 10 days of hospitalization for hepato-cutaneous fistula formation and tract epithelial maturation for the advancement of cholangioscope, which causes a significant financial burden as well as discomfort associated with fistula formation to the patients.

The SpyGlass™ DS Direct Visualization System (Boston Scientific Corp., Natick, Mass.) can be applied directly into the bile duct via the working channel of the duodenoscope. It can directly visualize the intra-ductal lesions with high-resolution digital imaging and it also has a working channel that allows the use of forcep, electrohydraulic lithotripsy (EHL) and Holmium Laser. So, it has the advantage of being able to directly examine intraductal lesions and perform treatment under the 'endoscopic view' which enables improved sensitivity of the diagnosis and the success rate of the treatment.

Intrahepatic duct (IHD) stone is difficult to treat by ERCP under fluoroscopy because IHD lesion is far from the orifice of bile duct (ampulla of Vater) and usually accompanied with IHD stenosis that causes technical difficulty. In addition, even if the stone is located in an extrahepatic bile duct (EHD; common hepatic duct and common bile duct), it is difficult to treat by ERCP in the case of a huge stone that has risk of incarceration. Therefore in these cases, bile duct stones have been being treated by PTCS. If the SpyGlass™ DS Direct Visualization System is used for the treatment of IHD/EHD stone that is not treatable with ERCP, it have potential benefits of reducing the financial burden and patient's discomfort caused by the PTCS significantly. Thus, we will investigate the usefulness of the SpyGlass™ DS Direct Visualization System for the treatment of IHD stones and huge EHD stones in terms of cost and success rate.

In this study, we will evaluate the treatment efficacy and cost-effectiveness of the SpyGlass™ DS Direct Visualization System facilitated management for IHD/EHD stones. The efficacy, cost-effectiveness and safety will be compared with historical cohort of percutaneous transhepatic cholangiography (PTCS)

ELIGIBILITY:
Inclusion Criteria:

1. IHD stones disease that cannot be treated with the ERCP.
2. Huge EHD stone disease that required mechanical/electrohydraulic lithotripsy, according to investigator's clinical decision.

Exclusion Criteria:

1. Patients who disagree with the study
2. Patients who underwent total gastrectomy
3. Patients with IHD stones located in a peripheral IHD where spyglass cannot reach

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Total hospital stay (# of days) | from admission to 1 month after discharge
  Total hospital day
Total procedure-related cost | from admission to 1 month after discharge
  Total cost from the date of admission and until date of first out-patient clinic follow-up

SECONDARY OUTCOMES:
Efficacy; Technical success rate | 1. after a month of ERCP procedure 2. after 3 months of ERCP procedure
  successful complete stone removal
Safety; Procedure-related complication rate | 1. after a month of ERCP procedure 2. after 3 months of ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: Moon Jae Chung, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No